CLINICAL TRIAL: NCT03372603
Title: A Placebo-controlled, Double-blind (Sponsor Open), Randomized, Crossover Study to Assess the Efficacy, Safety, and Tolerability of GSK2798745 in Participants With Chronic Cough
Brief Title: A Study to Assess the Effectiveness and Side Effects of GSK2798745 in Participants With Chronic Cough
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study terminated due to lack of efficacy of GSK2798745 in chronic cough.
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 207702; 2017-002265-21 (EudraCT Number)
Record Dates: First submitted 2017-12-08; First posted 2017-12-13 (Actual); Results first posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-08

CONDITIONS: Cough
Keywords: GSK2798745, efficacy, safety, chronic cough, crossover study
MeSH Terms: conditions — Cough; Chronic Cough | interventions — GSK2798745

STUDY DESIGN:
Intervention Model Description: This is a multi-center, randomized, placebo-controlled, double-blind, two-period crossover study. Each subject will be screened (screening may be conducted across more than 1 visit); each subject will have 2 treatment periods (each 7 days) with a washout period of 14 to 21 days between the treatment periods; and each subject will have a follow-up visit (within 7 to 10 days after their last dose). Each subject will be involved in the study for a maximum of 10 and a half weeks.
Who Masked: Participant, Investigator
Masking Description: All study staff involved in clinical assessments (which includes the investigator, sub-investigators, other site staff), and the subject will be blinded to the treatment allocated to individual subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence AB (Experimental): Subjects will receive GSK2798745 matching placebo tablets (two tablets on Day 1 followed by one tablet once daily for 6 days), via oral route (treatment period of total 7 days). After a washout period of 14 to 21 days, subjects will then receive 4.8 mg (two tablets of 2.4 mg) GSK2798745 on Day 1, followed by 2.4 mg GSK2798745 tablets once daily for 6 days via oral route (treatment period of total 7 days).
  Interventions: Drug: GSK2798745; Drug: Placebo
- Treatment Sequence BA (Experimental): Subjects will receive 4.8 mg (two tablets of 2.4 mg) GSK2798745 on Day 1, followed by 2.4 mg GSK2798745 tablets once daily for 6 days via oral route (treatment period of total 7 days). After a washout period of 14 to 21 days, subjects will then receive GSK2798745 matching placebo tablets (two tablets on Day 1 followed by one tablet once daily for 6 days), via oral route (treatment period of total 7 days).
  Interventions: Drug: GSK2798745; Drug: Placebo

INTERVENTIONS:
Drug: GSK2798745 — GSK2798745 tablets will be available as white to almost white, round, film-coated tablets (micronized active pharmaceutical ingredient [API]) to be taken with a glass of water (approximately 240 mL).
Drug: Placebo — Placebo tablets will be available as white to almost white, round, film-coated tablets to be taken with a glass of water (approximately 240 mL).

SUMMARY:
GSK2798745 is a potent and selective transient receptor potential vanilloid 4 (TRPV4) channel blocker being investigated for the treatment of chronic cough. This is a multi-center, randomized, placebo-controlled, double-blind, two-period crossover study with a purpose to evaluate efficacy and safety of GSK2798745. Each subject will have 2 treatment periods, and will be randomized to one of the following treatments in each period: A) Placebo matching to GSK2798745 once daily for 7 days. B) 4.8 milligrams (mg) GSK2798745 on Day 1, followed by 2.4 mg GSK2798745 once daily for 6 days. There will be a washout period of 14 to 21 days between the treatment periods. A maximum of 48 subjects will be enrolled in the study and the total duration of participation in the study will be maximum of 10 and a half weeks including follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years of age inclusive, at the time of signing the informed consent.
* Chronic idiopathic cough for >=1 year (before screening), defined as: a cough that is unresponsive to at least 8 weeks of targeted treatment, or a cough for which no objective evidence of an underlying trigger has been determined, despite medical investigations.
* No significant findings on chest imaging (chest X-ray [CXR] or Computed tomography scan) within 12 months before screening (subjects with an abnormal CXR within 12 months, from a temporary process, will be allowed to participate if a repeat CXR is normal).
* Forced expiratory volume in one second (FEV1) >=80% of the predicted normal value (at screening), or documented evidence of FEV1 >=80% within the 6 months before screening.
* Score of >=40 millimeters (mm) on the Cough Severity Visual Analogue Scale (VAS) at Screening.
* Body weight >=50 kilogram (kg) and body mass index (BMI) within the range 18 to 40 kilogram per meter square (kg/m^2) (inclusive) at screening.
* A male participant must agree to follow the contraception requirements stated in the protocol from the time of first dose of study treatment until 2 weeks after last dose of study treatment, and refrain from donating sperm during this period.
* A female participant is eligible to participate if she is not of childbearing potential.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* History or current evidence of any serious or clinically significant gastrointestinal, renal, endocrine, neurologic, hematologic or other condition that is uncontrolled on permitted therapies or that would, in the opinion of the investigator or the medical monitor, make the subject unsuitable for inclusion in this study.
* History or current evidence of chronic productive cough.
* History of acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting within the 6 months before screening.
* Active ulcer disease or gastrointestinal bleeding at the time of screening (positive fecal occult blood test [FOBT] at screening).
* History of stroke or seizure disorder within 5 years of screening.
* Respiratory tract infection within 6 weeks of screening.
* Subject who, in the investigator's opinion, poses a significant suicide risk. Evidence of serious suicide risk may include any history of suicidal behavior and/or any evidence of suicidal ideation on any questionnaires e.g. Type 4 or 5 on the Columbia Suicidality Severity Rating Scale (C-SSRS) in the last 6 months (assessed at screening).
* Alanine transferase (ALT) > twice the upper limit of normal (ULN) at screening.
* Bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%) at screening.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QT interval corrected (QTc) >450 milliseconds (msec) or QTc >480 msec in subjects with bundle branch block at screening.
* Use of a listed prohibited medication within the restricted timeframe relative to the first dose of study treatment.
* Use of a strong inhibitors or inducers of cytochrome P450 (CYP) 3A or pglycoprotein.
* Participation in the study would result in loss of blood or blood products in excess of 500 milliliters (mL) within 3 months of screening.
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Current enrollment or past participation within the 3 months before screening in any clinical study involving an investigational study treatment or any other type of medical research.
* Positive human immunodeficiency virus (HIV) antibody test at screening.
* Presence of Hepatitis B surface antigen (HBsAg) at screening.
* Positive Hepatitis C antibody test result at screening or within 3 months prior to starting study treatment.
* Positive Hepatitis C ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study treatment.
* Cardiac troponin at screening > ULN for the assay.
* History of alcohol abuse within 6 months of screening, in the opinion of the investigator.
* Current smoker or history of smoking within the 6 months before screening, or a cumulative history of >= 20 pack years. Pack years = (Number of cigarettes smoked/day/20) x (Number of years smoked)
* Sensitivity to any of the study treatments, or components thereof, or drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2018-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (4):
- United Kingdom (4):
  - GSK Investigational Site, Manchester, Lancashire
  - GSK Investigational Site, Belfast
  - GSK Investigational Site, Cottingham
  - GSK Investigational Site, North Shields

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 4 centers in the United Kingdom. Participants who met eligibility criteria entered a 2-period crossover study. Participants were randomized to either placebo or GSK2798745 in each Treatment Period (each 7 days, with a 14-21 day washout). Total duration of participation was 10.5 weeks. Study terminated on grounds of futility
Pre-assignment Details: A total of 34 participants were screened of which 17 failed screening and 17 participants were included in the study.
Groups:
- Placebo/GSK2798745: Participants were administered two tablets of placebo on Day 1 followed by one tablet of placebo on Days 2 to 7 of treatment period 1. In treatment period 2, participants received two tablets of 2.4 milligrams (mg) GSK2798745 each on Day 1 followed by one tablet of 2.4 mg GSK2798745 on Days 2 to 7. All doses were administered once daily via the oral route with a glass of water. The treatment periods were separated by a wash-out period of 14 to 21 days.
- GSK2798745/Placebo: Participants were administered two tablets of 2.4 mg GSK2798745 on Day 1 followed by one tablet of 2.4 mg GSK2798745 on Days 2 to 7 of treatment period 1. In treatment period 2, participants received two tablets of placebo on Day 1 followed by one tablet of placebo on Days 2 to 7. All doses were administered once daily via the oral route with a glass of water. The treatment periods were separated by a wash-out period of 14 to 21 days.
Period: Treatment Period 1 (Up to 7 Days)
Arm/Group | Placebo/GSK2798745 | GSK2798745/Placebo
Started | 9 | 8
Completed | 9 | 8
Not Completed | 0 | 0
Period: Wash-out Period (14-21 Days)
Arm/Group | Placebo/GSK2798745 | GSK2798745/Placebo
Started | 9 | 8
Completed | 8 | 8
Not Completed | 1 | 0
Not completed — Sponsor terminated study treatment | 1 | 0
Period: Treatment Period 2 (Up to 7 Days)
Arm/Group | Placebo/GSK2798745 | GSK2798745/Placebo
Started | 8 | 8
Completed | 7 | 8
Not Completed | 1 | 0
Not completed — Study closed/Terminated | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All participants who were randomized to either of the two treatment sequences Placebo/GSK2798745 and GSK2798745/Placebo and received GSK2798745 and placebo in either Treatment period 1 or 2 were included. All doses were administered once daily via the oral route with a glass of water. The treatment periods were separated by a wash-out period of 14 to 21 days.
Arm/Group | All Study Participants
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.0 (9.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 2
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian-Japanese/East Asian (EA)/South EA Heritage | 1
  White | 16

OUTCOME MEASURES:

1. Primary Outcome: Total Cough Counts During Day Time Hours Following 7-days of Dosing
Description: Coughs were monitored using the VitaloJAK cough monitor. The total cough counts during day-time (10 hours) was calculated from the time of the monitor being attached i.e. immediately after dosing on Day 7 to 10 hours past the time of monitoring. Total cough counts were log-transformed prior to analysis. A non-informative prior was used. Analysis was performed using a Bayesian mixed model adjusting for subject-level and period-adjusted baselines, treatment and period. Subject-level baseline is defined as the mean of the two period-specific baselines. Period-adjusted baseline is defined as the difference between the period-specific baseline and subject-level baseline for each period. Posterior median and 95% credible interval is reported. All Subjects Population included all randomized participants who took at least 1 dose of study treatment. Participants were analyzed according to the treatment they actually received.
Time Frame: Up to 10 hours post-dose on Day 7 of each treatment period
Population: All Subjects Population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (95% Confidence Interval); unit: Cough counts
Groups:
- Placebo: Participants were administered two tablets of placebo on Day 1 followed by one tablet of placebo on Days 2 to 7 in either treatment period 1 or 2. All doses were administered once daily via the oral route with a glass of water. The treatment periods were separated by a wash-out period of 14 to 21 days.
- GSK2798745: Participants were administered two tablets of 2.4 mg GSK2798745 on Day 1 followed by one tablet of 2.4 mg GSK2798745 on Days 2 to 7 in either treatment period 1 or 2. All doses were administered once daily via the oral route with a glass of water. The treatment periods were separated by a wash-out period of 14 to 21 days.
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 17 | 15
Cough counts | 180.570 [137.852 to 235.446] | 241.105 [181.383 to 320.600]
Statistical Analysis 1: Comparison: Placebo vs GSK2798745; Test type: Other; Ratio = 1.336, 90% CI 2-sided [0.965 to 1.847] — Treatment comparison ratio of GSK2798745 and placebo using posterior median ratio and 90% credible interval is presented

2. Secondary Outcome: Number of Participants Reporting Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, associated with liver injury and impaired liver function or any other situations as per medical or scientific judgment.
Time Frame: Up to 45 days
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 17 | 16
Participants
  Any AE | 9 | 11
  Any SAE | 0 | 0

3. Secondary Outcome: Change From Baseline Values for Clinical Chemistry Parameters: Alkaline Phosphatase (ALP), Alanine Aminotransferase (ALT), Aspartate Amino Transferase (AST) and Creatinine Kinase (CK)
Description: Blood samples were collected for the analysis of clinical chemistry parameters including ALP, ALT, AST and CK. Baseline was defined as latest pre-dose assessment with a non-missing value in each treatment period. Change from Baseline was calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and Day 8 of each treatment period
Population: All Subjects Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 17 | 14
International units per liter
  ALP | 1.8 (9.28) | -3.1 (6.75)
  ALT | 0.2 (2.31) | -0.2 (5.32)
  AST | -0.6 (3.69) | -0.5 (2.65)
  CK | -3.0 (21.71) | -12.1 (52.12)

4. Secondary Outcome: Change From Baseline Values for Clinical Chemistry Parameter: Direct Bilirubin, Total Bilirubin and Creatinine
Description: Blood samples were collected for the analysis of clinical chemistry parameters including direct bilirubin, total bilirubin and creatinine. Baseline was defined as latest pre-dose assessment with a non-missing value in each treatment period. Change from Baseline was calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and Day 8 for each treatment period
Population: All Subjects Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 17 | 14
Micromoles per liter
  Direct bilirubin | 0.1 (1.11) | 0.0 (0.78)
  Total bilirubin | -0.4 (3.41) | -0.4 (3.25)
  Creatinine | 0.31 (6.458) | 1.70 (4.031)

5. Secondary Outcome: Change From Baseline Values for Clinical Chemistry Parameters: Calcium, Glucose, Potassium, Sodium and Urea
Description: Blood samples were collected for the analysis of clinical chemistry parameters including calcium, glucose, potassium, sodium and urea/blood urea nitrogen (BUN). Baseline was defined as latest pre-dose assessment with a non-missing value in each treatment period. Change from Baseline was calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and Day 8 of each treatment period
Population: All Subjects Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 17 | 14
Millimoles per liter
  Calcium | 0.011 (0.0588) | 0.019 (0.0782)
  Glucose | -0.22 (1.234) | -0.06 (0.956)
  Potassium | 0.09 (0.299) | 0.09 (0.270)
  Sodium | 0.2 (1.44) | -0.1 (1.46)
  Urea | 0.18 (0.683) | -0.36 (0.908)

6. Secondary Outcome: Change From Baseline Values for Clinical Chemistry Parameter: Total Protein
Description: Blood samples were collected for the analysis of clinical chemistry parameter total protein. Baseline was defined as latest pre-dose assessment with a non-missing value in each treatment period. Change from Baseline was calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and Day 8 of each treatment period
Population: All Subjects Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 17 | 14
Grams per liter | 1.2 (2.65) | 0.9 (2.53)

7. Secondary Outcome: Number of Participants With Abnormal Values of Cardiac Troponin
Description: Cardiac troponin values was measured in participants.
Time Frame: Up to 45 days
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 17 | 16
Participants | NA — Not applicable (NA) indicates Troponin I values were recorded as less than lower limit of quantification (<0.02) at all time points. | NA — NA indicates Troponin I values were recorded as less than lower limit of quantification (<0.02) at all time points.

8. Secondary Outcome: Change From Baseline Values for Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Total Neutrophils, Platelet Count and White Blood Cell (WBC) Count
Description: Blood samples were collected for the analysis of hematology parameters including basophils, eosinophils, lymphocytes, monocytes, total neutrophils, platelet count and WBC count. Baseline was defined as latest pre-dose assessment with a non-missing value in each treatment period. Change from Baseline was calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and Day 8 of each treatment period
Population: All Subjects Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Giga units per liter
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 17 | 15
Giga units per liter
  Basophils | 0.005 (0.0250) | -0.005 (0.0316)
  Eosinophils | -0.005 (0.0400) | -0.007 (0.0758)
  Lymphocytes | 0.019 (0.3065) | -0.002 (0.2608)
  Monocytes | -0.012 (0.1110) | 0.027 (0.1012)
  Total neutrophils | 0.186 (0.5817) | 0.064 (1.0102)
  Platelet count | 6.8 (13.57) | 6.9 (19.76)
  WBC count | 0.20 (0.614) | 0.09 (1.276)

9. Secondary Outcome: Change From Baseline Values for Hematology Parameter: Hemoglobin
Description: Blood samples were collected for the analysis of hematology parameter: hemoglobin. Baseline was defined as latest pre-dose assessment with a non-missing value in each treatment period. Change from Baseline was calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and Day 8 for each treatment period
Population: All Subjects Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 17 | 15
Grams per liter | 0.5 (2.29) | 0.5 (3.52)

10. Secondary Outcome: Change From Baseline Values for Hematology Parameter: Hematocrit
Description: Blood samples were collected for the analysis of hematology parameter: hematocrit. Baseline was defined as latest pre-dose assessment with a non-missing value in each treatment period. Change from Baseline was calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and Day 8 of each treatment period
Population: All Subjects Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 17 | 15
Percentage of red blood cells in blood | 0.0020 (0.01009) | 0.0029 (0.00979)

11. Secondary Outcome: Change From Baseline Values for Hematology Parameter: Mean Corpuscular Hemoglobin (MCH)
Description: Blood samples were collected for the analysis of hematology parameter: MCH. Baseline was defined as latest pre-dose assessment with a non-missing value in each treatment period. Change from Baseline was calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and Day 8 for each treatment period
Population: All Subjects Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 17 | 15
Picograms | -0.07 (0.377) | -0.09 (0.442)

12. Secondary Outcome: Change From Baseline Values for Hematology Parameter: Mean Corpuscular Volume (MCV)
Description: Blood samples were collected for the analysis of hematology parameter: MCV. Baseline was defined as latest pre-dose assessment with a non-missing value in each treatment period. Change from Baseline was calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and Day 8 of each treatment period
Population: All Subjects Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 17 | 15
Femtoliters | -0.1 (2.01) | -0.1 (1.53)

13. Secondary Outcome: Change From Baseline Values for Hematology Parameter: Red Blood Cell (RBC) Count
Description: Blood samples were collected for the analysis of hematology parameter: RBC count. Baseline was defined as latest pre-dose assessment with a non-missing value in each treatment period. Change from Baseline was calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and Day 8 for each treatment period
Population: All Subjects Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Tera units per liter
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 17 | 15
Tera units per liter | 0.04 (0.112) | 0.03 (0.103)

14. Secondary Outcome: Change From Baseline Values for Hematology Parameter: Reticulocytes
Description: Blood samples were collected for the analysis of hematology parameter: reticulocytes. Baseline was defined as latest pre-dose assessment with a non-missing value in each treatment period. Change from Baseline was calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and Day 8 for each treatment period
Population: All Subjects Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of reticulocytes in blood
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 17 | 15
Percentage of reticulocytes in blood | -0.0002 (0.00300) | -0.0002 (0.00260)

15. Secondary Outcome: Number of Participants With Abnormal Urinalysis Data
Description: Urine samples were collected for analysis of urinalysis data by dipstick method. Number of participants with abnormal urinalysis data has been presented. Abnormality was defined as value of potential clinical importance (PCI). PCI was flagged when a result changed from negative on Day 1 (pre-dose) to positive on Day 8.
Time Frame: Up to Day 8
Population: All Subjects Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 17 | 15
Participants | 4 | 2

16. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: Blood pressure was measured at indicated time points in supine position after 5 minutes rest for the participant. Baseline was defined as latest pre-dose assessment with a non-missing value in each treatment period. Change from Baseline was calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (pre-dose on Day 1) and Day 8 of each treatment period
Population: All Subjects Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 17 | 15
Millimeters of mercury
  DBP | -0.2 (8.59) | -0.5 (13.07)
  SBP | 1.6 (12.65) | 0.9 (20.10)

17. Secondary Outcome: Change From Baseline in Temperature
Description: Temperature was measured at indicated time points in supine position after 5 minutes rest for the participant. Baseline was defined as latest pre-dose assessment with a non-missing value in each treatment period. Change from Baseline was calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (pre-dose on Day 1) and Day 8 of each treatment period
Population: All Subjects Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 17 | 15
Degrees Celsius | 0.02 (0.635) | -0.05 (0.331)

18. Secondary Outcome: Change From Baseline in Heart Rate
Description: Heart rate was measured at indicated time points in supine position after 5 minutes rest for the participant. Baseline was defined as latest pre-dose assessment with a non-missing value in each treatment period. Change from Baseline was calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (pre-dose on Day 1) and Day 8 of each treatment period
Population: All Subjects Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 17 | 15
Beats per minute | 0.6 (8.65) | -1.3 (12.09)

19. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: Twelve-lead ECG was obtained using an ECG machine that automatically calculated the heart rate and measured PR, QRS, QT, and corrected QT (QTc) intervals. Number of participants with abnormal-clinically significant and abnormal-not clinically significant values has been presented.
Time Frame: Baseline (pre-dose on Day 1) and Day 8 of each treatment period
Population: All Subjects Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category title).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2798745
Number analyzed (Participants) | 17 | 16
Participants
  Day 1 pre-dose, not clinically significant,n=17,16 | 2 | 1
  Day 1 pre-dose, clinically significant, n=17,16 | 0 | 0
  Day 8, not clinically significant, n=17,15: number analyzed (Participants) | 17 | 15
  Day 8, not clinically significant, n=17,15 | 2 | 1
  Day 8, clinically significant, n=17,15: number analyzed (Participants) | 17 | 15
  Day 8, clinically significant, n=17,15 | 0 | 1

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from the start of the treatment up to 45 days
Description: AEs and SAEs were collected for All Subjects population
Arm/Group | Placebo | GSK2798745
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 9/17 | 11/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=17) | GSK2798745 (N=16)
Headache (Nervous system disorders) | 3 (3) | 7 (7)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 2 (2)
Feeling cold (General disorders) | 1 (1) | 0 (0)
Suprapubic pain (General disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 1 (1) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/03/NCT03372603/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-07): https://cdn.clinicaltrials.gov/large-docs/03/NCT03372603/SAP_001.pdf